CLINICAL TRIAL: NCT05016232
Title: Developing and Pilot Testing an Adaptive Intervention to Facilitate PrEP Uptake and Maximize PrEP Adherence Among At-Risk Transgender Women
Brief Title: Adaptive Intervention to Facilitate PrEP Uptake/Adherence Among Transgender Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Matthew Mimiaga, ScD, MPH, MA, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH122499-01A1 (NIH)
Record Dates: First submitted 2021-08-09; First posted 2021-08-23 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Prevention
Keywords: Transgender women (TGW); HIV Prevention; PrEP
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength Based Case Management (SBCM) & PrEP adherence training and counseling (Experimental): Stage 1: Support, facilitate, and assist in linkage to PrEP clinic and to facilitate initiation of, and obtaining, PrEP medications.
  Stage 2: Stepped Intervention:
  1. Initially TGW in this arm will receive daily 2-way gender-affirming text message reminders, and
  2. Then those continuing to have poor adherence will receive the 4 (once per week for 3 to 4 weeks) more intensive counseling session with a clinical interventionist.
  Interventions: Behavioral: PrEP N' Shine: Strength Based Case Management (Stage 1); Behavioral: PrEP N' Shine: Stepped Adherence Training and Counseling (Stage 2)
- Standard of Care:Stage 1 and Stage 2 (No Intervention): Stage 1: Referral to local PrEP clinic Stage 2: Standard clinical PrEP care: Doctor visit every three months to assess for side effects, do blood work, and receive a HIV test.

INTERVENTIONS:
Behavioral: PrEP N' Shine: Strength Based Case Management (Stage 1) — Support, facilitate, and assist in linkage to PrEP clinic and to facilitate initiation of, and obtaining, PrEP medications.
  Arms: Strength Based Case Management (SBCM) & PrEP adherence training and counseling
Behavioral: PrEP N' Shine: Stepped Adherence Training and Counseling (Stage 2) — 1. Initially TGW in this arm will receive daily 2-way gender-affirming text message reminders, and
  2. Then those continuing to have poor adherence will receive the 4 (once per week for 3 to 4 weeks) more intensive counseling session with a clinical interventionist.
  Arms: Strength Based Case Management (SBCM) & PrEP adherence training and counseling

SUMMARY:
"PrEP N' Shine" is a two-stage randomized controlled pilot trial which utilizes a behavioral intervention to optimize the uptake and adherence of Pre-exposure Prophylaxis (PrEP) in Transgender women (TGW).

DETAILED DESCRIPTION:
The "PrEP N' Shine" package includes two behavioral intervention components:

1. Peer-led, strengths-based case management (SBCM) for PrEP linkage and uptake, and
2. A resource-efficient, adaptive "stepped-care" technology and counseling intervention that addresses individualized barriers to optimal use.

Stage 1: TGW will be equally randomized to receive either the strengths-based case management or standard of care referral to PrEP clinic.

Stage 2: Those from stage 1 who initiate PrEP , regardless of stage 1 randomization condition, will then be equally randomized to either the "PrEP N' Shine" adherence intervention or standard of care comparison condition.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or older
* Male sex at birth
* Self-identify as a woman, a transgender woman, or another identity along the male-to-female gender spectrum
* PrEP naïve
* PrEP indicated per CDC guidelines (incl. HIV negative)
* Owns a cell phone or willing to use one in the study
* Able to understand and speak English or Spanish

Exclusion Criteria:

* Unable to provide informed consent due to severe mental or physical illness, cognitive impairment, or substance intoxication at time of visit
* Has lived in RI for less than three months (as a means to enhance participant retention)
* Discovery of active suicidal ideation or major mental illness (e.g. untreated psychosis or mania) at the time of interview (these patients will be referred immediately for treatment, but may join the study when this is resolved)
* Laboratory or clinical findings that would preclude PrEP initiation (e.g. Hepatitis B infection, decreased creatinine clearance)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Must self-identify as a woman, a transgender woman, or another identity along the male-to-female gender spectrum
Enrollment: 123 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Verified medical visit and PrEP prescription | Stage 1: one month post-baseline
  Linkage to care and PrEP Initiation measured through verified medical appointment at PrEP Clinic and pharmacy through medical release.
Concentrations of TFV-DP in Dried Blood Spots at 3 months | Stage 2: 3 months post-baseline
  Dried Blood Spots (DBS) to be sent to the laboratory to test for tenofovir-diphosphate (700+ fmol/punch - corresponding to levels that are consistent with taking 4+ pills per week), which will serve as a biological measure of PrEP adherence.
Concentrations of TFV-DP in Dried Blood Spots at 6 months | Stage 2: 6 months post-baseline
  Dried Blood Spots (DBS) to be sent to the laboratory to test for tenofovir-diphosphate (700+ fmol/punch - corresponding to levels that are consistent with taking 4+ pills per week), which will serve as a biological measure of PrEP adherence

SECONDARY OUTCOMES:
Change in sexual risk behavior based on self report | Stage 2: Change from baseline sexual risk behavior at 6 months
  Change in sexual risk behavior to be measured using AIDS-Risk Behavior Assessment (ARBA), a computerized self-interview designed to assess self-reported sexual behaviors. Sexual risk questions refer to three types of sexual behavior (anal, oral, vaginal) and assess detailed sexual risk information by partner type (transactional, casual, main) and by HIV-status, whether protected or unprotected, and whether in the context of substance use in past 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Mimiaga, ScD, MPH, MA, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for LGBTQ+ Advocacy, Research & Health, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that this data will be presented annually on data collected after the second year when sufficient baseline data is collected. It is anticipated that most of the papers and data-based projects/presentations will happen in year 3, when all of the baseline data is collected, and the 3 month outcome has occurred for all participants. Sharing of the findings will involve a primary paper describing the study outcome and a paper that describes the intervention, as well as submitting to lead workshops on the intervention approach at relevant national meetings and conferences. Raw data for additional analysis will be available to outside individuals through contacting the MPIs. Information regarding the availability of data for analysis will be listed on the MPIs' web pages. Contact information for the MPIs will be listed in all manuscripts and publications as another means to access data.